CLINICAL TRIAL: NCT00844168
Title: Phase I Adjuvant Trial of Sorafenib in Hepatocellular Carcinoma Patients After Liver Transplantation
Brief Title: Sorafenib Tosylate in Treating Patients With Liver Cancer Who Have Undergone a Liver Transplant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6697; NCI-2009-01659 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Adult Primary Hepatocellular Carcinoma; Advanced Adult Primary Liver Cancer; Localized Resectable Adult Primary Liver Cancer; Localized Unresectable Adult Primary Liver Cancer; Recurrent Adult Primary Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (adjuvant sorafenib tosylate after liver transplant) (Experimental): Patients receive sorafenib tosylate PO twice daily on days 1-28. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sorafenib tosylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: sorafenib tosylate — Given orally
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of sorafenib tosylate in treating patients with liver cancer who have undergone a liver transplant. Sorafenib tosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving sorafenib after liver transplant may be an effective treatment for liver cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Establish the safety and toxicity profile of sorafenib administered daily to hepatocellular carcinoma (HCC) patients who have undergone orthotopic liver transplantation.

SECONDARY OBJECTIVES:

I. Determine explant and allograft expression of vascular endothelial growth factor (VEGF), platelet derived growth factor receptor (PDGFR), microvessel density (CD34) and Ki67 (proliferation marker).

OUTLINE: Patients receive sorafenib tosylate orally (PO) twice daily on days 1-28. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years, and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HCC on explant, who have not received prior systemic anti-cancer treatment for HCC
* HCC patients who have undergone orthotopic liver transplantation, are at high risk for tumor recurrence or who have high suspicion or documentation of tumor recurrence
* Patients who have a life expectancy of at least 12 weeks
* Patients must have one of the following disease states:

  * Patients are 4 weeks beyond and less than 60 days from liver transplant surgery (to first study treatment) who have no residual hepatocellular carcinoma following liver transplantation;
  * Patients with post transplant recurrent hepatocellular carcinoma within the liver or at an extra hepatic site, diagnosed by radiographic imaging (computed tomography [CT] or magnetic resonance imaging [MRI]) consistent with hepatocellular carcinoma or proved by biopsy, within 24 months of transplantation;
  * Post-transplant patients with rising alpha-feta protein level > 500ng/mL, even in the absence of confirmed disease within 24 months of transplant
* Patients must have one of the following explant histological features of HCC:bilobar tumor; macrovascular invasion; or multifocality; if patients have well-differentiated HCC, they must have all three features
* Patients who have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Platelet count >= 60 x 10^9/L
* Hemoglobin >= 8.5 g/dL
* Total bilirubin =< 3 mg/dL
* Alanine transaminase (ALT) and aspartate transaminase (AST) =< 5 x upper limit of normal
* Amylase and lipase =< 1.5 x the upper limit of normal
* Serum creatinine =< 1.5 x the upper limit of normal
* Prothrombin time (PT)-international normalized ratio (INR) =< 2.3 or PT 6seconds above control
* Patients who give written informed consent

Exclusion Criteria:

* Previous or concurrent cancer that is distinct in primary site or histology from HCC, EXCEPT cervical carcinoma in situ, treated basal cell carcinoma,superficial bladder tumors (Ta, Tis & T1); any cancer curatively treated > 3 years prior to entry is permitted
* Renal failure requiring hemo- or peritoneal dialysis
* History of cardiac disease: congestive heart failure > New York Heart Association (NYHA) class 2; active coronary artery disease (CAD); cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers ordigoxin; or uncontrolled hypertension; myocardial infarction more than 6months prior to study entry is permitted
* Active clinically serious infections > grade 2 (National Cancer Institute -Common Terminology Criteria for Adverse Events version 3.0)
* Known history of human immunodeficiency virus (HIV) infection
* Known central nervous system tumors including metastatic brain disease
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Known or suspected allergy to the investigational agent or any agent given in association with this trial
* Patients unable to swallow oral medications
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study
* Pregnant or breast-feeding patients; women of childbearing potential must have a negative pregnancy test performed within seven days prior to the start of study drug; both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial
* Prior use of any systemic anti-cancer chemotherapy for HCC
* Prior use of systemic investigational agents for HCC
* Prior use of Raf-kinase inhibitors (RKI), VEGF inhibitors, MEK inhibitors or Farnesyl transferase inhibitors
* Use of biologic response modifiers, such as granulocyte colony-stimulating factor (G-CSF), within 3 weeks prior to study entry (G-CSF and other hematopoietic growth factors may be used in the management of acute toxicity, such as febrile neutropenia, when clinically indicated or at the discretion of the investigator; however, they may not be substituted for a required dose reduction)
* Patients taking chronic erythropoietin are permitted provided no dose adjustment is undertaken within 1 month prior to the study or during the study
* Autologous bone marrow transplant or stem cell rescue within four months of start of study drug
* Concomitant treatment with rifampin and St John's wort
* Concomitant anti-coagulation therapy with warfarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-01; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) as defined by the Common Terminology for Adverse Events (CTAE) version 3 | 28 days
  Defined as grade >= 3 nonhematologic/hematologic toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Edward Lin, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States